CLINICAL TRIAL: NCT07106814
Title: Safety and Efficacy of Metabolically Armed Tumor-lnfiltrating Lymphocytes (Meta10-TIL) for the Treatment of Advanced Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Collaborators: Leman Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: META10-TIL-09
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumors
Keywords: Meta10-TIL; Advanced solid tumors; Liver cancer; Cervical cancer; IL-2
MeSH Terms: conditions — Liver Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of Metabolically Armed tumor-infiltrating lymphocytes(Meta10-TIL) (Experimental): Patients will receive a nonmyeloablative lymphodepletion chemotherapy with cyclophosphamide and fludarabine before TIL cells infusion.Meta10-TIL cells will be infused on day 0.
  Interventions: Drug: Metabolically Armed TIL cells

INTERVENTIONS:
Drug: Metabolically Armed TIL cells — Each subject receive metabolically armed TIL cells by intravenous infusion.
  Other Names: Meta10-TIL

SUMMARY:
A Study of Metabolically Armed Tumor-Infiltrating Lymphocytes (Meta10-TIL) Therapy for Patients With Advanced Solid Tumors

DETAILED DESCRIPTION:
This is an open-label study. This study is indicated for advanced solid tumors. The selections of dose levels and the number of subjects are based on clinical trials of similar products and the outcomes of our preliminary clinical studies.

1. Main research objectives:

   To evaluate the safety of metabolically armed tumor-infiltrating lymphocytes (TILs) in patients with advanced solid tumors.
2. Secondary research objectives:

(1)To evaluate the objective response rate (ORR),duration of response (DOR), progression-free survival (PFS), and disease control rate (DCR) of metabolically armed tumor-infiltrating lymphocytes (Meta10-TIL) with RECIST V1.1; (2) To evaluate the overall survival (OS); (3) Characterize the pharmacokinetic (PK) and pharmacodynamic (PD) profiles of Meta10-TILs.

ELIGIBILITY:
Inclusion Criteria:

* The patient or his/her guardian voluntarily signed the informed consent;
* Age >18 years and ≤70 years, male or female;
* Patients with advanced solid tumors who have been confirmed by histopathology or cytology and have received at least first-line of treatment:

  1. Recurrent/metastatic/persistent (persistent defined as disease progression after initial treatment) cervical cancer, including squamous cell carcinoma (SCC), adenosquamous carcinoma (ASC), and adenocarcinoma (AC), and not eligible for curative surgery and/or radiotherapy:

     1. Recurrent/metastatic/persistent cervical cancer with prior failure (disease progression or intolerable toxicity) of at least 1 but no more than 3 systemic therapies;
     2. Systemic therapy is defined as any chemotherapy or multi-drug combination chemotherapy regimen recommended by guidelines used for cervical cancer;
     3. Chemotherapy or chemoradiotherapy administered as neoadjuvant or adjuvant therapy is not counted as a prior line of systemic therapy.
  2. Or, classified as Stage Ⅳ cervical cancer according to the International Federation of Gynecology and Obstetrics (FIGO 2018) staging criteria (studies have shown that patients with early-stage cancer may have better outcomes after TIL therapy. After confirming significantly superior efficacy compared to marketed TIL products, researchers can relax staging criteria according to their judgment);
  3. Histologically or cytologically confirmed locally advanced/metastatic liver malignancies (including hepatocellular carcinoma, intrahepatic cholangiocarcinoma, and metastatic liver cancer):

     1. For hepatocellular carcinoma (HCC), classified as Barcelona Clinic Liver Cancer (BCLC) Stage C or Stage B unsuitable for local therapy or progressed after local therapy;
     2. For locally advanced liver cancer, patients must have failed at least first-line systemic therapies recommended by guidelines (disease progression or intolerable toxicity);
     3. Unresectable intrahepatic cholangiocarcinoma patients must have failed at least 1 but no more than 3 prior systemic therapies recommended by guidelines(disease progression or intolerable toxicity);
     4. Metastatic liver cancer ineligible for curative surgery based on primary tumor TNM (Tumor Node Metastasis) staging; for metastatic liver cancer, patients must have failed at least 2 but no more than 3 guideline-recommended systemic therapies (disease progression or intolerable toxicity);
     5. Liver function Child-Pugh score ≤7;
     6. Or patients deemed by the investigator to be unsuitable for existing standard treatments, or who refuse standard therapy.
  4. Advanced solid tumors that have progressed after prior standard therapy or are intolerant to toxicity, for which no standard treatment options are currently available, or for other reasons cannot receive the current standard treatment, including but not limited to primary or metastatic triple-negative breast cancer (TNBC), non-small cell lung cancer (NSCLC) (excluding neuroendocrine tumors or mixed types with >10% neuroendocrine components), ovarian cancer (OC), head and neck cancer (HNC), and colorectal cancer (CRC).
* The subject has residual lesions suitable for surgical resection (≥1.5 cm) or biopsy (core needle biopsy specimens: ≥4 passes with 16G needle or ≥6 passes with 18G needle) to generate tumor-infiltrating lymphocytes (TILs). For cervical cancer subjects, tumor tissue meeting either ≥0.5 cm in diameter or ≥400 mm³ in volume is acceptable. Fresh tumor tissue for TIL production should preferably be obtained from proximal metastatic lymph nodes or the periphery of tumor lesions. The sampled lesion has not received local therapy (e.g., radiotherapy, radiofrequency ablation, oncolytic virus, etc.) or such interventions have occurred ≥3 months prior and the lesion has progressed after local treatment;
* Expected life expectancy ≥3 months;
* After tumor resection/puncture, the subject must have at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1) for efficacy evaluation;
* Eastern Cooperative Oncology Group (ECOG) performance status was 0-1 (subjects with stable brain metastases require investigator assessment);
* Adequate organ function:

  1. Hematological (no transfusions, platelet infusions, or growth factor support [except recombinant erythropoietin] within 7 days prior to enrollment):

     1. Absolute neutrophil count (ANC)≥1x10^9/L;
     2. Platelet count (PLT) ≥80 × 10^9/L;
     3. Hemoglobin (Hb) ≥90.0 g/L;
  2. Blood chemistry:

     1. Estimated creatinine clearance ≥40 mL/min (calculated by Cockcroft-Gault formula);
     2. Alanine aminotransferase (ALT) ≤3 × upper limit of normal (ULN);
     3. Aspartate aminotransferase (AST) ≤3 × ULN;
     4. Total bilirubin (TBIL) ≤2 mg/dL (subjects with Gilbert-Meulengracht syndrome ≤3 mg/dL);
     5. Serum AST and ALT ≤5 × ULN (subjects with liver metastasis);
  3. Adequate pulmonary reserve defined as ≤Grade 1 dyspnea and oxygen saturation >91% on room air;
  4. Left ventricular ejection fraction (LVEF) ≥45% by echocardiography or multigated acquisition (MUGA) scan, with hemodynamic stability;
* In the investigator's judgment, the subject must have recovered from prior anticancer therapy toxicities to Grade 1 or lower (except for specific Grade 2 or lower toxicities deemed irreversible in a short period of time as judged by the investigator, e.g., alopecia) and be eligible for preconditioning chemotherapy and TIL therapy;
* Subjects with documented ≥Grade 2 diarrhea or colitis from prior immune checkpoint inhibitor therapy must be asymptomatic for ≥6 months before tumor resection, with normal colonoscopy (visual assessment) post-immunotherapy (excluding colorectal cancer patients);
* Subjects with immune-related endocrinopathies (e.g., hypothyroidism) may enroll if stable for ≥6 weeks and controlled with hormone replacement therapy (non-corticosteroid);
* Women of childbearing potential and all male subjects must agree to use highly effective methods of contraception at the time of informed consent, and continue within 1 year after Meta10-TILs infusion.

Exclusion Criteria:

* Presence of bone metastases only.
* Active central nervous system (CNS) metastases (except for stable brain metastases not requiring medication or steroid dependence for ≥3 months).
* Use of Chinese herbal medicine or botanical drugs with antitumor indications within 1 week before preconditioning.
* Systemic corticosteroid therapy (≥10 mg/day prednisone or equivalent) or other immunosuppressive drugs within 2 weeks before preconditioning (excluding inhaled, topical, or physiological replacement therapy).
* Subjects who have undergone major surgery within 4 weeks before enrollment (as assessed by the investigator) or planned major surgery during the study (excluding scheduled surgery for Meta10-TILs preparation); Major surgery refers to Grade 3 & 4 surgeries as defined by China's Administrative Measures for Clinical Application of Medical Technology (effective on May 1, 2009).
* History of other malignancies within 3 years before screening or concurrent malignancies (except for locally treated malignancies with no recurrence risk for ≥1 year, e.g., non-melanoma skin cancer, bladder cancer).
* Any form of primary immunodeficiency disorder (e.g., severe combined immunodeficiency [SCID] or acquired immunodeficiency syndrome [AIDS]).
* History of organ transplantation.
* Active hepatitis B (HBsAg positive or anti-HBc positive with HBV-DNA >1000 copies/mL) or hepatitis C (HCV-RNA positive).
* Anti-HIV antibody positive or anti-syphilis antibody positive.
* Uncontrolled acute life-threatening bacterial, viral, or fungal infections (e.g., positive blood culture ≤72 hours before Meta10-TILs infusion).
* Patients who have received a live or attenuated vaccination within 4 weeks before preconditioning.
* Unstable angina and/or myocardial infarction within 6 months before signing informed consent; Uncontrolled thrombotic events, severe bleeding, or deep vein thrombosis (DVT) within 12 months before signing informed consent.
* History of neurological or psychiatric disorders, including epilepsy or dementia.
* History of hypersensitivity to drugs (e.g., cyclophosphamide, fludarabine, IL-2, Meta10-TILs components, gentamicin, etc.).
* High bleeding risk per investigator assessment, including but not limited to: tumor encasement/infiltration of major blood vessels (e.g., carotid artery, jugular vein, bronchial artery); other high-risk features (e.g., fistula, cavitary lesions, history of previous bleeding [≤60 days]).
* Patients who have received other investigational therapies within 30 days before signing informed consent.
* Other conditions deemed ineligible for the study by the investigator (e.g., Grade ≥3 adverse events in previous immunotherapy).

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2027-08-15 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events(AEs) | 1 year post Meta10-TIL infusion
  To characterize the safety profile of Meta10-TIL in patients with advanced solid tumor as assessed by incidence of adverse events. Adverse events will be graded by the National Cancer Institute Common Terminology Criteria for Adverse Events(NCI CTCAE) version 5.0.

SECONDARY OUTCOMES:
Objective response rate(ORR) | 1 year post Meta10-TIL infusion
  To evaluate the proportion of participants who have a confirmed partial response (PR) and complete response (CR) per RECIST v1.1 as assessed by the investigator.
Overall survival(OS) | 1year post Meta10-TIL infusion
  OS is measured from the date of the infusion of Meta10-TIL to the date of the subjects' death.
Duration of Response(DOR) | 1 year post Meta10-TIL infusion
  To evaluate the duration from the time that criteria are met for CR or PR per RECIST v1.1 as assessed by the investigator until disease progression or death due to any cause.
Progression-free survival(PFS) | 1 year post Meta10-TIL infusion
  The time from the start of Meta10-TIL treatment for the subjects to the first disease progression or death for any reason.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Provincial Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No